CLINICAL TRIAL: NCT04783155
Title: Effect of Inspiratory Muscle Training on Physiological Function and Clinical Outcomes After Lung Transplant: A Randomized Controlled Trial
Brief Title: Effect of Inspiratory Muscle Training on Physiological Function and Clinical Outcomes After Lung Transplant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bryan Taylor, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20-012778
Record Dates: First submitted 2021-02-22; First posted 2021-03-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Post-Lung Transplantation Bronchiectasis
Keywords: Inspiratory muscle training; post lung transplant; exercise capacity; breathing
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-blinded, randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 12-weeks pulmonary rehabilitation training plus inspiratory muscle training (Experimental): To assess maximum inspiratory pressure, you will be asked to breathe through a device called POWERBreathe Plus®. This device is commercially available and will be provided to you by the study. You will be asked to use this device twice per day, 5 days per week, for 12 weeks. Each session will require you to breathe into the device 30 times. You can use the device at home.
  Interventions: Device: POWERBreathe Plus®; Other: Cardiopulmonary rehabilitation post lung transplant
- 12-weeks pulmonary rehabilitation plus placebo (inactive) inspiratory muscle (Placebo Comparator): To assess maximum inspiratory pressure with placebo, you will be asked to breathe through a device called POWERBreathe Plus®. This device is commercially available and will be provided to you by the study. You will be asked to use this device twice per day, 5 days per week, for 12 weeks. Each session will require you to breathe into the device 30 times. You can use the device at home. The resistance will be set to about 5% throughout the study.
  Interventions: Device: POWERBreathe Plus®; Other: Cardiopulmonary rehabilitation post lung transplant

INTERVENTIONS:
Device: POWERBreathe Plus® — Commercially available pressure-threshold device
Other: Cardiopulmonary rehabilitation post lung transplant — Pulmonary function, lung diffusing capacity for carbon monoxide, inspiratory muscle strength, and diaphragm dimensions will be assessed in each patient. Each patient will also undergo a cardiopulmonary exercise test (CPET), 6 minute walk test, and an inspiratory muscle endurance test

SUMMARY:
The purpose of this research is to study the effect of training the inspiratory muscles (i.e. the muscle that allow you to breath-in) on exercise capacity, quality of life, and short-term clinical outcomes in patients post lung transplant.

ELIGIBILITY:
Inclusion Criteria:

- All patients who undergo single- or double-lung transplant at Mayo Clinic Florida.

Exclusion Criteria:

* Patients who do not survive the intra-operative period during the transplant surgery.
* Patients undergoing retransplantation.
* Patients undergoing multiorgan transplantation.
* Patients who are not willing to or who are unable to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Maximal inspiratory mouth pressure (MIP) measured in cmH2O | 12 weeks
  The maximal strength generating capacity of the inspiratory muscles.

SECONDARY OUTCOMES:
Maximal oxygen uptake (V̇O2max) measured in mL/kg/min | 12 weeks
  Vo2 max is the maximal measured oxygen uptake during a symptom limited exercise test.

OTHER OUTCOMES:
Six-minute walk test distance (6MWTd) measured in meters (m) | 12 weeks
  Distance walked during a 6 minute test
Peak work rate (Wpeak) (watts) | 12 weeks
  The maximal work achieved in watts during a symptom limited exercise test.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Taylor, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials